CLINICAL TRIAL: NCT01461759
Title: A Phase II Trial of Docetaxel / Cisplatin in Patients With Recurrent or Stage IVb Endometrial Cancer
Brief Title: Efficacy Study of Chemotherapy to Treat Advanced or Recurrent Endometrial Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Asan Medical Center (Other)
Collaborators: Boryung Pharmaceutical Co., Ltd (Industry)
Responsible Party: Principal Investigator, Joo-Hyun Nam, Professor, Asan Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ANSGOG-002
Record Dates: First submitted 2011-10-25; First posted 2011-10-28 (Estimated); Last update posted 2017-05-31 (Actual); Status verified 2017-05

CONDITIONS: Advanced or Recurrent Endometrial Cancer
MeSH Terms: conditions — Endometrial Neoplasms | interventions — Cisplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Chemotherapy (Experimental): Docetaxel 70mg/m2BSA + Cisplatin 60mg/m2BSA, q 3 weeks, 8cycles
  Interventions: Drug: Doctaxel; Drug: Cisplatin

INTERVENTIONS:
Drug: Doctaxel — Docetaxel 70mg/m2BSA, q 3 weeks, 8 cycles
Drug: Cisplatin — Cisplatin 60mg/m2BAS, q 3 weeks, 8 cycles

SUMMARY:
The purpose of this study is to treat advanced or recurrent endometrial cancer, paclitaxel-containing regimen is the preferred chemotherapeutic regimen which is selected by most physicians. Docetaxel may have similar efficacy and more favorable treatment related toxicity profile as tested in epithelial ovarian cancer trials. Therefore, the investigators aimed to evaluate the efficacy and safety of docetaxel plus cisplatin in patients with advanced or recurrent endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed chemotherapy naïve endometrial cancer
* One of following histology Endometrioid, UPSC, CCCa, squamous, adenosquamous, mixed
* FIGO stage IVb or recurrent endometrial cancer (incurable by surgery and/or RT)
* At least one measurable lesion by RECIST on CT
* ECOG PS: 0-2
* Age: 20-75
* Adequate organ function BM: ANC≥1,000/mm3, Plt≥100X103/mm3 Kidney: Creatinine<1.25 × UNL이고, GFR ≥ 60 Liver: AST, ALT< 3×UNL, T- bil<1.5 mg/ mm3
* Informed Consent
* Contraception during study period

Exclusion Criteria:

* Previous chemotherapy
* RT, hormone therapy, or immunotherapy within 1 month
* Other malignant disease
* Uncontrolled medical disease
* Infection requiring antibiotics
* Symptomatic CHF, RF, Angina, Arrhythmia, etc.
* Neurosis or psychosis
* Pregnancy, breast-feeding
* Etc.

Ages: 20 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 59 (Estimated)
Dates: Start 2011-10; Primary Completion 2017-12 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Response rate | 3 months after completion of study treatment

SECONDARY OUTCOMES:
Progression-free survival | 2 years after completion of study treatment
Number of Participants with Adverse Events as a Measure of Safety and Tolerability | Before each chemotherapy, an expected average of 3 weeks
Quality of life | 3 months after completion of study treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Asan Medical Center, Seoul, South Korea